CLINICAL TRIAL: NCT04871581
Title: Adjunctive Treatment of Chronic Migraine Using an Oral Dental Device: Overview and Results of a Placebo-Controlled Crossover Study
Brief Title: Adjunctive Treatment of Chronic Migraine Using an Oral Dental Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChairsideSplint.com (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NTI v Placebo
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Chronic Migraine, Headache
Keywords: single blinded study
MeSH Terms: conditions — Headache

STUDY DESIGN:
Intervention Model Description: Single blinded cross-over study
Who Masked: Participant
Masking Description: Participants were advised that two different designs of device were being compared to each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Device (Active Comparator): Subjects receiving the FDA-cleared device
  Interventions: Device: NTI-tss
- Placebo (Placebo Comparator): Subjects receiving the sham device
  Interventions: Device: Placebo

INTERVENTIONS:
Device: NTI-tss — FDA cleared device for prophylactic treatment of medically diagnosed migraine pain
  Arms: Device
Device: Placebo — Similar to Device, but having no influence on clenching intensity
  Arms: Placebo

SUMMARY:
Single blinding study comparing FDA cleared device for prevention of medically diagnosed migraine pain to placebo.

DETAILED DESCRIPTION:
In order to determine if nocturnal jaw clenching can be an influence on chronic migraine pain, the FDA cleared "NTI" (Nociceptive Trigeminal Inhibition) device with the Indications for Use of "for prophylactic treatment of medically diagnosed migraine pain" was compared to a similar device that had no influence on jaw clenching.The HIT-6 (Headache Impact Test) score was selected as the outcome measure, as the goal was to focus on improving disability in sufferer's lives, as in chronic migraine, changes in headache days may not be as helpful as improving disability.

ELIGIBILITY:
Inclusion Criteria: Diagnosed with chronic migraine at a neurology clinic -

Exclusion Criteria: none

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Improvement of negative impact on life | one month
  At least a one-category improvement in subject's HIT-6 score

CONTACTS AND LOCATIONS:
Locations (1):
- Boyd James, Solana Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silberstein SD, Lipton RB. Chronic daily headache. Curr Opin Neurol. 2000 Jun;13(3):277-83. doi: 10.1097/00019052-200006000-00008. PMID 10871251
- [Background] Pascual J, Colas R, Castillo J. Epidemiology of chronic daily headache. Curr Pain Headache Rep. 2001 Dec;5(6):529-36. doi: 10.1007/s11916-001-0070-6. PMID 11676887
- [Background] Rozen TD. Migraine prevention: what patients want from medication and their physicians (a headache specialty clinic perspective). Headache. 2006 May;46(5):750-3. doi: 10.1111/j.1526-4610.2006.00429.x. PMID 16643577
- [Background] Goadsby PJ. Migraine pathophysiology. Headache. 2005 Apr;45 Suppl 1:S14-24. doi: 10.1111/j.1526-4610.2005.4501003.x. PMID 15833086
- [Background] Graff-Radford SB, Newman AC. The role of temporomandibular disorders and cervical dysfunction in tension-type headache. Curr Pain Headache Rep. 2002 Oct;6(5):387-91. doi: 10.1007/s11916-002-0081-y. PMID 12207852
- [Background] Steele JG, Lamey PJ, Sharkey SW, Smith GM. Occlusal abnormalities, pericranial muscle and joint tenderness and tooth wear in a group of migraine patients. J Oral Rehabil. 1991 Sep;18(5):453-8. doi: 10.1111/j.1365-2842.1991.tb01690.x. PMID 1800695
- [Background] Lamey PJ, Barclay SC. Clinical effectiveness of occlusal splint therapy in patients with classical migraine. Scott Med J. 1987 Feb;32(1):11-2. doi: 10.1177/003693308703200105. PMID 3563468
- [Background] Clark GT, Sakai S, Merrill R, Flack VF, McArthur D, McCreary C. Waking and sleeping temporalis EMG levels in tension-type headache patients. J Orofac Pain. 1997 Fall;11(4):298-306. PMID 9656905
- [Background] Graff-Radford SB. Oromandibular disorders and headache. A critical appraisal. Neurol Clin. 1990 Nov;8(4):929-45. PMID 2259320
- [Background] Yap AU, Chua AP. Sleep bruxism: Current knowledge and contemporary management. J Conserv Dent. 2016 Sep-Oct;19(5):383-9. doi: 10.4103/0972-0707.190007. PMID 27656052
- [Background] Burnett CA, Fartash L, Murray B, Lamey PJ. Masseter and temporalis muscle EMG levels and bite force in migraineurs. Headache. 2000 Nov-Dec;40(10):813-7. doi: 10.1046/j.1526-4610.2000.00147.x. PMID 11135025
- [Background] Chandu A, Suvinen TI, Reade PC, Borromeo GL. The effect of an interocclusal appliance on bite force and masseter electromyography in asymptomatic subjects and patients with temporomandibular pain and dysfunction. J Oral Rehabil. 2004 Jun;31(6):530-7. doi: 10.1111/j.1365-2842.2004.01377.x. PMID 15189309
- [Background] Nishigawa K, Bando E, Nakano M. Quantitative study of bite force during sleep associated bruxism. J Oral Rehabil. 2001 May;28(5):485-91. doi: 10.1046/j.1365-2842.2001.00692.x. PMID 11380790
- [Result] Castillo J, Munoz P, Guitera V, Pascual J. Kaplan Award 1998. Epidemiology of chronic daily headache in the general population. Headache. 1999 Mar;39(3):190-6. doi: 10.1046/j.1526-4610.1999.3903190.x. PMID 15613213
- [Derived] Blumenfeld AM, Boyd JP. Adjunctive treatment of chronic migraine using an oral dental device: overview and results of a randomized placebo-controlled crossover study. BMC Neurol. 2022 Mar 4;22(1):72. doi: 10.1186/s12883-022-02591-8. PMID 35246048